CLINICAL TRIAL: NCT01006057
Title: A Trial Investigating the Pharmacokinetic and Safety of NN1250 in Subjects With Various Degrees of Renal Impairment and in Subjects With Normal Renal Function
Brief Title: A Trial Investigating the NN1250 Concentration-time Curve in Subjects With Various Degrees of Renal Impairment and in Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-1990; 2009-009466-14 (EudraCT Number); U1111-1111-0810 (Other: WHO)
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- ESRD (Experimental)
  Interventions: Drug: insulin degludec
- Mild (Experimental)
  Interventions: Drug: insulin degludec
- Moderate (Experimental)
  Interventions: Drug: insulin degludec
- Normal (Experimental)
  Interventions: Drug: insulin degludec
- Severe (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Single dose of 0.4 U/kg body weight injected s.c. (under the skin) in subjects with end stage renal disease
  Arms: ESRD
Drug: insulin degludec — Single dose of 0.4 U/kg body weight injected s.c. (under the skin) in subjects with mild renal impairment
  Arms: Mild
Drug: insulin degludec — Single dose of 0.4 U/kg body weight injected s.c. (under the skin) in subjects with moderate renal impairment
  Arms: Moderate
Drug: insulin degludec — Single dose of 0.4 U/kg body weight injected s.c. (under the skin) in healthy volunteers
  Arms: Normal
Drug: insulin degludec — Single dose of 0.4 U/kg body weight injected s.c. (under the skin) in subjects with severe renal impairment
  Arms: Severe

SUMMARY:
This trial was conducted in Europe. The aim of this clinical trial was to evaluate if the NN1250 (insulin degludec/insulin 454) concentration-time curve is altered to such an extent that the dose should be adjusted in subjects with impaired renal function compared to the dose for subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Subject with normal renal function or renal impairment (mild, moderate, severe or end stage renal disease (ESRD) requiring haemodialysis)
* Body mass index maximum 40.0 kg/m^2

Exclusion Criteria:

* Subject with any disease or condition which the Investigator feels would interfere with the trial except for conditions associated with renal impairment in the group of subjects with compromised renal function. Diabetes mellitus can be accepted in the group of patients with renal impairment, but not in subjects with normal renal function
* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Significant history of alcoholism or drug/chemical abuse
* Not able or willing to refrain from smoking during the inpatient period

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Area under the insulin degludec concentration-time curve | from 0 to 120 hours after trial product administration

SECONDARY OUTCOMES:
Maximum observed insulin degludec concentration | from 0 to 120 hours after trial product administration
Renal clearance of insulin degludec after single-dose | from 0 to 24 hours after trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Budapest, Hungary

REFERENCES:
- [Result] Kiss I, Arold G, Roepstorff C, Bottcher SG, Klim S, Haahr H. Insulin degludec: pharmacokinetics in patients with renal impairment. Clin Pharmacokinet. 2014 Feb;53(2):175-83. doi: 10.1007/s40262-013-0113-2. PMID 24163264
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com